CLINICAL TRIAL: NCT02322333
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of MLD10 in the Prevention of Migraine Headache in Adults
Brief Title: MLD10 in the Prevention of Migraine in Adults
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pharmalyte Solutions LLC (Industry)
Collaborators: Clinvest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MLD10-002
Record Dates: First submitted 2014-12-17; First posted 2014-12-23 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Magnesium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MLD10 (Active Comparator): Subjects randomized to MLD10 will be dispensed a 28 day supply of magnesium L-lactate dehydrate for daily treatment. A total of 120 caplets will be given each time at Visit 2, 3, and 4. Additional overage will be given to account for the 3 day window. Subjects will be instructed to take two caplets of study medication BID (twice a day) at about the same time each day. Subjects will be instructed regarding storage requirements and will be asked to return all used/partially used/unused medication containers at the next office visit.
  Interventions: Drug: MLD10
- Placebo (Placebo Comparator): Subjects randomized to placebo will be dispensed a 28 day supply of matching placebo for daily treatment. A total of 120 caplets will be given each time at Visit 2, 3, and 4. Additional overage will be given to account for the 3 day window. Subjects will be instructed to take two caplets of study medication BID (twice a day) at about the same time each day. Subjects will be instructed regarding storage requirements and will be asked to return all used/partially used/unused medication containers at the next office visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MLD10
  Other Names: elemental magnesium
  Arms: MLD10
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled, randomized, multi-center study. Subjects agreeing to participate in the study and meet the entry criteria assessed at the screening visit, will begin a 28 day baseline period to confirm their diagnosis, as well as establish baseline migraine characteristics. During this baseline period, subjects will continue treating their migraines as usual, simply recording the information in a daily headache diary. Subjects who, after completing the baseline, continue to meet entrance criteria will be eligible to enter into the treatment phase and be randomized according to the Clinvest generated randomization schedule. Approximately 142 subjects (71 subjects per arm) will be randomized and enter the treatment phase receiving MLD10 or placebo in a 1:1 design at 6 United States sites. Diary assessments will collect study medication adherence, pain severity, headache symptoms, acute medication usage, and unusual symptoms. Serum samples will be collected and analyzed for ionized magnesium, electrolytes, and creatinine.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized, placebo-controlled, parallel study of MLD10 for the prevention of migraine headache. The study population will consist of approximately 142 male and female subjects between 18 and 65 years of age with frequent episodic migraine as defined by International Classification of Headache Disorders-3beta criteria. Two MLD10 (243 mg (milligrams) of elemental magnesium) or placebo caplets will be taken twice daily for a total daily dose of 486 mg.

VISIT 1 - SCREENING

The following will be completed at Visit 1:

1. Obtain written Informed Consent. The informed consent will be obtained in accordance with Good Clinical Practices (GCP) and all applicable regulatory requirements from each subject prior to participation in the study.
2. Verify Inclusion/Exclusion Criteria. Subjects will meet all the inclusion and none of the exclusion criteria.
3. Obtain demographics (race, ethnicity, sex, date of birth)
4. Obtain medical, medication, and headache history. Data collected will include medical history and diagnoses, age at onset of migraine and other pertinent migraine/headache history, history of acute and prophylactic headache medications within the past 30 days, and history of other recent/concomitant medications.
5. Obtain date of last menstrual cycle and perform urine pregnancy test, if appropriate. Results of the pregnancy test must be negative to continue in study.
6. Perform physical and neurological examinations.
7. Measure vital signs (height, weight, resting heart rate, and blood pressure).
8. Review Baseline Headache Diary. Subjects will be instructed to complete a daily online headache diary. Assessments to be captured are start/stop time, severity, associated symptoms, use of rescue medications, and unusual symptoms.
9. Administer Columbia-Suicide Severity Rating Scale (C-SSRS).
10. Schedule Visit 2.

VISIT 2 - RANDOMIZATION

1. Verify Inclusion/Exclusion Criteria. Subjects must continue to meet all inclusion (including ≥ 3 days of migraine during baseline) and none of the exclusion criteria.
2. Perform urine pregnancy test, if appropriate. Results of the pregnancy test must be negative to continue in study.
3. Measure vital signs (weight, resting heart rate, and blood pressure).
4. Record any changes to concomitant medications.
5. Record any Serious Adverse Events (SAE) since signing the Informed Consent.
6. Review Baseline Headache Diary for completeness and continuing eligibility.
7. Randomize subject
8. Review Month 1 Headache Diary instructions (same instructions as those discussed for Baseline Headache Diary).
9. Dispense Month 1 study medication. Subjects will be instructed how to take study medication, prohibited medications/foods, dosage limitations of study medication, and storage requirements. Subjects will be instructed to return all used/partially used/unused study medication at next office visit and medications reconciliation will be performed to ensure a compliance of at least 80%. Subjects not complying at an 80% level will be withdrawn, unless otherwise approved by the Sponsor and/or Clinvest. (Estimated to be < 10%)
10. Administer C-SSRS.
11. Administer MIDAS.
12. Collect serum samples for electrolytes, creatinine, and ionized Mg.
13. Schedule Visit 3.

VISIT 3 - END OF TREATMENT PERIOD MONTH 1

1. Record any changes to concomitant medications.
2. Record any Non-Serious Adverse Events (NSAE) and/or SAEs.
3. Perform urine pregnancy test, if appropriate. Results of the pregnancy test must be negative to continue in study.
4. Measure vital signs (weight, resting heart rate, and blood pressure).
5. Review Month 1 Headache Diary for completeness.
6. Review instructions for Month 2 Headache Diary (same instructions as those discussed for Month 1 Headache Diary).
7. Collect Month 1 unused study medication and used packaging. Confirm 85% compliance of medication usage per study protocol.
8. Dispense Month 2 study medication and review the dosage limitations of study medication, storage requirements, and to return all used/partially used/unused study medication at next office visit.
9. Perform drug accountability.
10. Administer C-SSRS.
11. Collect serum samples for electrolytes, creatinine, and ionized Mg.
12. Schedule Visit 4.

VISIT 4 - END OF TREATMENT PERIOD MONTH 2

1. Record any changes to concomitant medications.
2. Record any NSAEs/SAEs.
3. Perform urine pregnancy test, if appropriate. Results of the pregnancy test must be negative to continue in study.
4. Measure vital signs (weight, resting heart rate, and blood pressure).
5. Review Month 2 Headache Diary for completeness.
6. Review instructions for Month 3 Headache Diary (same instructions as those discussed for Month 2 Headache Diary).
7. Collect Month 2 unused study medication and used packaging. Confirm 85% compliance for medication usage per study protocol.
8. Dispense Month 3 study medication and review the dosage limitations of study medication, storage requirements, and to return all used/partially used/unused study medication at next office visit.
9. Perform drug accountability.
10. Administer C-SSRS.
11. Collect serum samples for electrolytes, creatinine, and ionized Mg.
12. Schedule Visit 5.

VISIT 5 - END OF TREATMENT PERIOD MONTH 3

1. Record any changes to concomitant medications.
2. Record any NSAEs/SAEs.
3. Perform urine pregnancy test, if appropriate.
4. Measure vital signs (weight, resting heart rate, and blood pressure)
5. Perform physical/neurological examinations.
6. Collect Month 4 unused study medication and used packaging.
7. Perform drug accountability.
8. Administer SGIC & complete PGIC.
9. Administer MIDAS.
10. Administer C-SSRS.
11. Collect serum samples for electrolytes, creatinine, and ionized Mg.
12. Exit subject.

ELIGIBILITY:
Inclusion Criteria:

1. male or female, in otherwise good health, 18 to 65 years of age.
2. history of frequent episodic migraine (3-14 migraine days per month) (with or without aura) according to the International Classification of Headache Disorders-3beta for at least 3 months.
3. onset of migraine before age 50.
4. stable history of migraine at least 3 months prior to screening.
5. not currently taking a migraine preventive or has been taking preventive for at least 30 days prior to screening and agrees to not start, stop, or change medication and/or dosage during the study period.
6. if female of childbearing potential, has a negative urine pregnancy test at Visits 1-5 and uses, or agrees to use, for the duration of the study, a medically acceptable form of contraception as listed:

   * complete abstinence from intercourse from 2 weeks prior to administration of study drug, throughout the study, and for 7 days after completion or premature discontinuation from the study; surgically sterile (hysterectomy or tubal ligation or otherwise incapable of pregnancy); sterilization of male partner when in a monogamous relationship; intrauterine device with published data showing lowest expected failure rate is less than 1% per year; double barrier method (i.e., 2 physical barriers OR 1 physical barrier plus spermicide) for a least 1 month prior to Visit 1 and throughout study; or hormonal contraceptives for at least 3 months prior to Visit 1 and throughout study.
7. completion of online diary must be ≥ 80% compliance, unless otherwise approved by the Sponsor and/or Clinvest.

Exclusion Criteria:

1. unable to understand the study requirements, the informed consent, or complete headache records as required per protocol.
2. pregnant, actively trying to become pregnant, or breast-feeding.
3. diagnosed with International Classification of Headache Disorders-3beta criteria for Chronic Migraine within 3 months prior to screening, at the time of screening, and/or during the baseline period.
4. experienced the following migraine variants: basilar migraine, aura without headache, familial hemiplegic migraine, complicated migraine, ophthalmoplegic migraine and retinal migraine within the last year.
5. history of medication overuse headache (MOH) (Appendix II) in the 3 months prior to study enrollment or during the baseline phase.
6. history of medication overuse (MO) of ergotamines, triptans, opioids, analgesics, NSAIDS and combination therapies, as defined by ICHD-3beta criteria and/or MO during baseline period.
7. history of substance abuse and/or dependence, in the opinion of the Investigator.
8. history of impaired renal function that, in the investigator's opinion, contraindicates participation in this study.
9. unstable neurological condition or a significantly abnormal neurological examination with focal signs or signs of increased intracranial pressure.
10. suffers from a serious illness, or an unstable medical condition, one that could require hospitalization, or could increase the risk of adverse events.
11. has significant risk of suicide, defined as a "yes" answer to any of the following questions on the Columbia-Suicide Severity Rating Scale (C-SSRS), either at the screening visit (when assessing the prior 12 months) or at visit 2 (when assessing time since the screening visit):

    1. Questions 4 or 5 on the suicidal ideation section
    2. Any question on any item in the suicidal behavior section
12. any psychiatric disorder with psychotic features, and/or any other psychiatric disorder not stable or well controlled, that would interfere in their ability to complete study activities.
13. hypersensitivity, intolerance, or contraindication to the use of magnesium L-lactate dehydrate or any of its components.
14. received any investigational agents within 30 days prior to Visit 1.
15. plans to participate in another clinical study at any time during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - The Research Center of Southern California, Carlsbad, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Physician Associates of Florida Research Department, Oviedo, Florida
  - Dr. B. Abraham, P.C., Snellville, Georgia
  - Westside Family Medical Center, P.C., Kalamazoo, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research, LLC, Springfield, Missouri
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Nashville Neuroscience Group, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- MLD10: Subjects randomized to MLD10 will be dispensed a 28 day supply of magnesium L-lactate dehydrate for daily treatment. A total of 120 caplets will be given each time at Visit 2, 3, and 4. Additional overage will be given to account for the 3 day window. Subjects will be instructed to take two caplets of study medication BID (twice a day) at about the same time each day. Subjects will be instructed regarding storage requirements and will be asked to return all used/partially used/unused medication containers at the next office visit.
  MLD10
- Placebo: Subjects randomized to placebo will be dispensed a 28 day supply of matching placebo for daily treatment. A total of 120 caplets will be given each time at Visit 2, 3, and 4. Additional overage will be given to account for the 3 day window. Subjects will be instructed to take two caplets of study medication BID (twice a day) at about the same time each day. Subjects will be instructed regarding storage requirements and will be asked to return all used/partially used/unused medication containers at the next office visit.
  Placebo
Period: Overall Study
Arm/Group | MLD10 | Placebo
Started | 80 | 77
Completed | 63 | 61
Not Completed | 17 | 16

BASELINE CHARACTERISTICS:
Groups:
- MLD10: All study participants randomized to MLD10 arm
- Placebo: All study participants randomized to Placebo arm
- Total: Total of all reporting groups
Arm/Group | MLD10 | Placebo | Total
Number analyzed (Participants) | 80 | 77 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.35 (12.72) | 44.74 (11.41) | 43.01 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 69 | 140
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 77 | 74 | 151
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 16 | 21
  White | 68 | 58 | 126
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Migraine Headache Days
Description: Comparison of the mean change from baseline in the frequency of migraine headache days per 28-day period ending with the cessation of treatment period month 3 in subjects treated with MLD10 versus placebo.
  A migraine headache day will be defined as a calendar day (00:00 to 23:59) with 4 or more hours of migraine headache, fulfilling International Classification of Headache Disorders-3beta criteria, and/or any headache of any duration with the use of migraine-specific acute medications(s) (i.e. ergot alkaloids, ergot combinations, opioids, triptans, combination analgesics [simple analgesics combined with opioids or barbiturate with or without caffeine]).
Time Frame: Day 1(Screening) - Day 116 (Visit 5 End of Study)
Population: The modified intent-to-treat (mITT) population included all randomized subjects who received at least one dose of study drug and obtained at least one endpoint measurement after treating. The mITT population excluded 7 subjects from the MLD10 arm and 6 participants from the Placebo arm. Total mITT analysis population: MLD10 = 73, Placebo = 71.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MLD10 | Placebo
Number analyzed (Participants) | 73 | 71
Days
  Baseline | 7.12 (2.94) | 6.92 (2.71)
  Treatment Period 3 | 5.53 (4.43) | 4.79 (4.20)

2. Secondary Outcome: Headache Days
Description: Comparison of the change from baseline of subjects treated with MLD10 versus placebo in the frequency of headache days during the 3 month treatment period.
  A headache day will be defined as any day not classified as a migraine day, but recorded headache of any severity and/or duration.
Time Frame: Day 1(Screening) - Day 116 (Visit 5 End of Study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MLD10 | Placebo
Number analyzed (Participants) | 73 | 71
Days
  Baseline | 9.01 (3.16) | 9.20 (3.70)
  Treatment Period 3 | 6.89 (5.36) | 6.25 (4.81)

3. Secondary Outcome: Headache Duration
Description: Change from baseline (28 day period) in the total cumulative minutes of headache during each 28-day treatment period month 1, 2, & 3 in subjects treated with MLD10 versus placebo.
  All headaches and/or migraines will be including in this outcome analysis.
Time Frame: Day 1(Screening) - Day 116 (Visit 5 End of Study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | MLD10 | Placebo
Number analyzed (Participants) | 73 | 71
Minutes
  Baseline | 410.03 (182.26) | 396.48 (166.75)
  Treatment Period 1 | 430.88 (242.35) | 369.03 (188.78)
  Treatment Period 2 | 443.89 (233.60) | 364.21 (186.09)
  Treatment Period 3 | 429.26 (228.59) | 383.70 (204.06)

4. Secondary Outcome: Pain Severity
Description: Change from baseline (28 day period) in the average pain severity at time of onset compared to each 28-day treatment period month 1, 2, & 3 in subjects treated with MLD10 versus placebo. Headache pain severity was measured on a scale 1 = Mild, 2 = Moderate, 3 = Severe.
Time Frame: Day 1(Screening) - Day 116 (Visit 5 End of Study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MLD10 | Placebo
Number analyzed (Participants) | 73 | 71
units on a scale
  Baseline | 2.16 (0.50) | 2.06 (0.37)
  Treatment Period 1 | 2.07 (0.54) | 1.93 (0.49)
  Treatment Period 2 | 1.99 (0.54) | 1.85 (0.53)
  Treatment Period 3 | 2.01 (0.49) | 1.86 (0.57)

5. Secondary Outcome: Acute Medication Usage
Description: Change from baseline (28 day period) in the total number of acute headache pain medications used during each 28 day treatment period month 1, 2, & 3 in subjects treated with MLD10 versus placebo.
Time Frame: Day 1(Screening) - Day 116 (Visit 5 End of Study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Medications
Arm/Group | MLD10 | Placebo
Number analyzed (Participants) | 73 | 71
Medications
  Baseline | 11.67 (7.64) | 11.08 (6.10)
  Treatment Period 1 | 9.74 (8.15) | 8.13 (6.23)
  Treatment Period 2 | 9.12 (7.08) | 8.61 (8.38)
  Treatment Period 3 | 9.18 (8.40) | 8.25 (8.67)

6. Secondary Outcome: Migraine Disability Assessment Scale (MIDAS)
Description: Change from Visit 2 to Visit 5 in the total MIDAS score in subjects treated with MLD10 versus placebo.
  The MIDAS test determines how severely migraines affect daily functioning. The responses of a variety of questions will be scored according to the questionnaire's scoring guide. A total score will be calculated ranging from 0-93. A score of 0-5 indicates little or no disability, 6-10 mild disability, 11-20, moderate disability, 21+ severe disability.
Time Frame: Day 29 (Randomization) & Day 116 (Visit 5 End of Study)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MLD10 | Placebo
Number analyzed (Participants) | 80 | 77
units on a scale
  Visit 2 | 33.94 (34.56) | 27.03 (25.41)
  Visit 5 | 27.14 (33.91) | 21.40 (18.64)

7. Secondary Outcome: Subject Global Impression of Change (SGIC)
Description: Comparison of SGIC at Visit 5 in subjects treated with MLD10 versus placebo.
  Global impression of change rated by the subject will be assessed using a 7-point Likert scale ranging from -3 to 3 with -3 = very much worse, -2 = much worse, -1 = minimally worse, 0 = no change, 1 = minimally improved, 2 = much improved, 3 = very much improved.
Time Frame: Day 116 (Visit 5 End of Study)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MLD10 | Placebo
Number analyzed (Participants) | 80 | 77
units on a scale | 1.25 (0.987) | 1.10 (1.23)

8. Secondary Outcome: Physician Global Impression of Change (PGIC)
Description: Comparison of PGIC at Visit 5 in subjects treated with MLD10 versus placebo.
  The PGIC will be an impression of change rated by the investigator using a 7-point Likert scale ranging from -3 to 3 with -3 = very much worse, -2 = much worse, -1 = minimally worse, 0 = no change, 1 = minimally improved, 2 = much improved, 3 = very much improved.
Time Frame: Day 116 (Visit 5 End of Study)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MLD10 | Placebo
Number analyzed (Participants) | 80 | 77
units on a scale | 1.07 (1.09) | 1.06 (1.12)

ADVERSE EVENTS:
Time Frame: Day 1 (Screening) - Day 116 (Visit 5 End of Study) for Serious Adverse Events Day 29 (Randomization) - Day 116 (Visit 5 End of Study) for Non-Serious Adverse Events
Groups:
- MLD10: All subjects randomized to MLD10 arm
- Placebo: All subjects randomized to Placebo arm
Arm/Group | MLD10 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/77
Serious Adverse Events (participants affected / at risk) | 1/80 | 1/77
Other Adverse Events (participants affected / at risk) | 17/80 | 15/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MLD10 (N=80) | Placebo (N=77)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MLD10 (N=80) | Placebo (N=77)
Diarrhoea (Gastrointestinal disorders) | 11 (12) | 5 (6)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Viral upper respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5)
Dizziness (Nervous system disorders) | 6 (8) | 1 (1)
Sinusitis (Infections and infestations) | 4 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-04-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT02322333/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT02322333/SAP_001.pdf